CLINICAL TRIAL: NCT04703543
Title: Pilot Study Evaluating the Role of Both PSMA and 64Cu-PET/CT Total Body in Patients With Locally Relapsed Prostate Cancer
Brief Title: Evaluating the Role of Both PSMA and 64Cu-PET/CT Total Body in Patients With Locally Relapsed Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Giuseppe Sanguineti, Professor, Regina Elena Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RS946/17(1974)
Record Dates: First submitted 2020-07-15; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Prostate Neoplasms
Keywords: PET-CT Scan; mpMRI; prostate neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: patients with metastatic prostatic cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pilot evaluation study on use PSMA and Cu-PET/CT — This study aims at assessing the detection rate of both PSMA and Cu-PET/CT on tissue relapse, study whether this method is equivalent to mpMR

SUMMARY:
The purpose of this study is to assess the detection rate of local relapse after radical prostatectomy with either PSMA or 64Cu-PET/CTs and whether the delineation of relapsed lesions using both methods can facilitate/change the therapeutic strategy of the radiation oncologist

DETAILED DESCRIPTION:
PET/TC is a diagnostic tool potentially able to detect, in a single session, both local and distant disease. However, the sensitivity of 18-F-PET/CT in the identification of relapse on the prostatic bed, varies greatly and depends on the value of PSA with which the examination is carried out, the size of the relapse in the lodge, the acquisition protocol and it is limited by the physiological hyperaccumulation of the tracer in the bladder. The sensitivity of 18F-Choline PET/TC in our hands is significantly higher than the one that is generally reported in the literature (76% with PSA values >1 ng/ml after radical prostatectomy), but still lower than the one of mpMR. PET/CT with 64Cu exceeds the limits of 18F-choline PET/TC in the study of the prostatic bed, as the tracer used (64Cu) is not excreted by urinary route and therefore does not accumulate in the bladder.

This study has the following objectives:

Primary objective: - To evaluate the detection rate of both 64Cu-PET/CT and PSMA-PET/CT of relapses in patients undergoing radical prostatectomy and subsequent biochemical recurrence;

Secondary objectives are:

* to assess any change in radiation therapy strategy in terms of lesion delineation and dose distribution at planning.
* to evaluate the performance of both methods (mpMR and PSMA/64Cu-PET/CT) in assessing the response to radiotherapy with or without androgen deprivation

ELIGIBILITY:
Criteria: Inclusion Criteria:

* Localized prostate adenocarcinoma (M0), any PSA value, any Gleason Score
* Previous radical surgery with subsequent undetectable PSA (<0.2 ng/ml)
* Biochemical recurrence (two consecutive PSA values of at least 0.2 ng/ml)
* M0 to 18F-choline PET/TC
* Local relapse at mpMR
* Age>18 years
* Performance Status 0-1 according to ECOG
* Informed written consent Exclusion Criteria:
* Detectable PSA after surgery
* Secondary bone lesions from prostate cancer or M1
* Hormone therapy started before staging examinations
* Previous pelvic radiotherapy
* Crohn's disease or ulcerative colitis (active phase)
* Psychiatric diseases
* Contraindication to MRI (metal prostheses, pacemakers, claustrophobia, etc.)
* Presence of coxo-femoral implants

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — prostatic neoplasm
Enrollment: 50 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
To calculate the detection rate of PSMA and Cu-PET/CT of relapses in patients undergoing radical prostatectomy and subsequent biochemical recurrence | 60 months
  Ratio between positive PSMA and Cu-PET/CT patients and the total of enrolled patients (positive MRI)

CONTACTS AND LOCATIONS:
Locations (1):
- Regina Elena National Cancer Institute, Rome, Italy

REFERENCES:
- [Derived] Bottero M, Faiella A, Giannarelli D, Farneti A, D'Urso P, Bertini L, Landoni V, Vici P, Sanguineti G. A prospective study assessing the pattern of response of local disease at DCE-MRI after salvage radiotherapy for prostate cancer. Clin Transl Radiat Oncol. 2022 Apr 27;35:21-26. doi: 10.1016/j.ctro.2022.04.010. eCollection 2022 Jul. PMID 35516461